CLINICAL TRIAL: NCT02367872
Title: Phase I Open-label, Parallel-group, Comparative Study to Evaluate the Effects of Renal or Hepatic Impairment on TAK-272 Pharmacokinetics With a Single Oral Administration of TAK-272 in Patients With Renal or Hepatic Impairment
Brief Title: Phase I Open-label Study to Evaluate Pharmacokinetics of TAK-272 in Participants With Renal or Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-272/CPH-012; U1111-1166-3774 (Registry Identifier: WHO); JapicCTI-152790 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Renal Impairment; Hepatic Impairment
Keywords: Drug therapy
MeSH Terms: conditions — Renal Insufficiency | interventions — imarikiren hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Participants with normal renal function: TAK-272 40 mg (Active Comparator): Fasted single oral administration of TAK-272 40 milligram (mg)
  Interventions: Drug: TAK-272
- Participants with mild renal impairment: TAK-272 40 mg (Experimental): Fasted single oral administration of TAK-272 40 mg
  Interventions: Drug: TAK-272
- Participants with moderate renal impairment: TAK-272 40 mg (Experimental): Fasted single oral administration of TAK-272 40 mg
  Interventions: Drug: TAK-272
- Participants with severe renal impairment: TAK-272 40 mg (Experimental): Fasted single oral administration of TAK-272 40 mg
  Interventions: Drug: TAK-272
- Hemodialysis participants: TAK-272 40 mg (Experimental): Fasted single oral administration of TAK-272 40 mg
  Interventions: Drug: TAK-272
- Participants with normal hepatic function: TAK-272 40 mg (Active Comparator): Fasted single oral administration of TAK-272 40 mg
  Interventions: Drug: TAK-272
- Participants with mild hepatic impairment: TAK-272 40 mg (Experimental): Fasted single oral administration of TAK-272 40 mg
  Interventions: Drug: TAK-272
- Participants with moderate hepatic impairment: TAK-272 40 mg (Experimental): Fasted single oral administration of TAK-272 40 mg
  Interventions: Drug: TAK-272

INTERVENTIONS:
Drug: TAK-272 — TAK-272 tablet

SUMMARY:
The purpose of this study is to examine the effects of renal and hepatic impairment on TAK-272 pharmacokinetics with a single oral administration of TAK-272 in participants with renal or hepatic impairment.

DETAILED DESCRIPTION:
This study is a phase I, open-label, parallel-group, comparative study to evaluate the effects of renal or hepatic impairment on pharmacokinetics of TAK-272 with a single oral administration of TAK-272 in participants with renal or hepatic impairment as compared with participants with normal renal and hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All participants

1. In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. Is either male or female and aged 20 to 85 years, inclusive, at the time of informed consent.
4. Weighs at least 45 kilogram (kg) for males and 40 kg for females and have a body mass index (BMI) of less than (<) 35.0 kilogram per square meter (kg/m^2) at screening and Day 1.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent until 12 weeks after study drug administration.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of informed consent until 1 month after the completion of the study.

   Participants with normal renal or hepatic function (Cohorts 1R and 1H)
7. Estimated glomerular filtration rate (eGFR) is greater than or equal to (>=) 90 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) at screening.
8. Based on the participant's medical history, clinical laboratory values, and physical examination findings, the investigator or subinvestigator judges the participant to be in good health (hypertension, type 2 diabetes, and hypercholesteremia or dyslipidemia are controlled, if present).
9. Is within +/-10 years of the mean age and +/-20 percent (%) of the mean weight for the 24 participants with renal impairment and 12 participants with hepatic impairment administered the study drug.

   Participants with renal impairment (Cohorts 2R, 3R, 4R, 5R)
10. Falls into any of the following categories:

    * With mild renal impairment (Cohort 2R): eGFR >=60 mL/min/1.73 m^2 and <90 mL/min/1.73 m^2 at screening.
    * With moderate renal impairment (Cohort 3R): eGFR >=30 mL/min/1.73 m^2 and <60 mL/min/1.73 m^2 at screening.
    * With severe renal impairment or end-stage renal failure (non-hemodialysis participants) (Cohort 4R): eGFR <30 mL/min/1.73 m^2 at screening.
    * Hemodialysis participants (Cohort 5R): with end-stage renal failure and little or no urine output who are undergoing hemodialysis 3 times weekly.
11. For non-hemodialysis participants, difference in eGFR obtained between 3 months and 7 days before screening from eGFR at screening is less than or equal to (<=) 30%.

    Participants with hepatic impairment (Cohorts 2H, 3H)
12. In observations during the screening period, those diagnosed with hepatic impairment corresponding to any of the following Child-Pugh classes:

    * With mild hepatic impairment (Cohort 2H): Child-Pugh class A.
    * With moderate hepatic impairment (Cohort 3H): Child-Pugh class B.
13. Is diagnosed by the investigator or subinvestigator with hepatic impairment that has remained stable during the 3 months before screening.

Exclusion Criteria:

All participants

1. Has received any investigational product within 16 weeks (112 days) prior to the start of study drug administration.
2. Has received TAK-272 in a previous clinical study.
3. Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. Has a history of cancer. This does not include individuals who have been in remission for at least 1 year prior to the start of screening and who are judged by the investigator or subinvestigator to have had no recurrence during the study.
5. Has a known hypersensitivity or allergy to any component of the TAK-272 formulation or renin inhibitors.
6. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
7. Has any positive urine drug test result at screening (including test for alcohol) if a non-hemodialysis participant.
8. Has taken any excluded medication or food product listed in the Excluded Medications and Dietary Products section during the period in which excluded medication use is prohibited, or needs to take any excluded medication or food product during the study.
9. Previously has undergone kidney or liver transplantation.
10. Has poor peripheral venous access.
11. Has undergone whole blood collection of 800 milliliter (mL) or more within 52 weeks (364 days) prior to the start of study drug administration.
12. Has undergone whole blood collection of 200 mL or more within 4 weeks (28 days) or 400 mL or more within 12 weeks (84 days) for males and 16 weeks (112 days) for females prior to the start of study drug administration.
13. Has undergone blood component collection within 2 weeks (14 days) prior to the start of study drug administration.
14. Has onset of myocardial infarction or coronary revascularization within 6 months before screening.
15. Has a history of abdominal surgery (excluding laparoscopic cholecystectomy or appendectomy without complications) or chest or non-peripheral vascular surgery within 6 months before screening.
16. Has onset of acute disease (example, renal and urinary tract disease) within 30 days before screening.
17. Has clinically significant abnormal electrocardiogram (ECG) in the screening period or the pretreatment examination.
18. Has clinically significant hyperkalemia.
19. If female, the participant is pregnant or lactating or intending to become pregnant before, during or within 1 month after participating in this study, or intending to donate ova during such time period.
20. If male, the participant intends to donate sperm during the course of this study or for 12 weeks thereafter.
21. In the opinion of the investigator or subinvestigator, is unlikely to comply with protocol or is unsuitable for any other reason.

    Participants with normal renal and hepatic function (Cohorts 1R and 1H)
22. Has uncontrolled, clinically significant hepatic, renal, neurologic, cardiovascular, blood, pulmonary, metabolic, gastrointestinal, urologic or endocrine disease, immune disease, infection or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
23. Has clinical laboratory results at screening suggestive of a clinically significant underlying disease other than controlled hypertension, type 2 diabetes, hypercholesteremia, or dyslipidemia.
24. Systolic blood pressure is <80 millimeter of mercury (mmHg) at screening, in the pretreatment examination, or in the examination prior to the start of study drug administration and has repeated instances of the findings listed below, suggesting the presence of hypotension:

    - Dizziness postural, facial pallor, cold sweats.
25. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is >2.0 times higher than the upper limit of normal at screening.
26. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, or serological reactions for syphilis at screening.

    Participants with renal impairment (Cohorts 2R, 3R, 4R, 5R)
27. Has uncontrolled, clinically significant hepatic, neurologic, cardiovascular, blood, pulmonary, metabolic, gastrointestinal, urologic or endocrine disease, immune disease, infection or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
28. Sitting systolic blood pressure is <110 mmHg at screening, in the pretreatment examination, or in the examination before administration on Day 1.
29. ALT or AST is >2.0 times higher than the upper limit of normal at screening.
30. Has a positive test result for HBsAg, HCV antibody, HIV antigen/antibody, or serological reactions for syphilis at screening.

    Participants with hepatic impairment (Cohorts 2H, 3H)
31. Has uncontrolled, clinically significant renal, neurologic, cardiovascular, blood, pulmonary, metabolic, gastrointestinal, urologic or endocrine disease, immune disease, infection or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
32. Has ascites requiring invasive treatment.
33. Systolic blood pressure is <80 mmHg at screening, in the pretreatment examination, or in the examination prior to the start of study drug administration and has repeated instances of the findings listed below, suggesting the presence of hypotension:

    - Dizziness postural, facial pallor, cold sweats.
34. eGFR is <60 mL/min/1.73 m^2 at screening.
35. Has a positive test result for HIV antigen/antibody or the participant has a positive test result for serological reactions for syphilis and syphilis is judged not to have been cured at screening.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (4):
- Japan (4):
  - Kurume, Fukuoka
  - Moriya, Ibaragi
  - Sagamihara, Kanagawa
  - Shinagawa, Tokyo

REFERENCES:
- [Derived] Shimasaki Y, Sakaki M, Itou M, Kobayashi T, Aso M, Kagawa T, Saiki T, Matsuno K, Sano Y, Shimizu K, Kuroda S, Koumura E. Pharmacokinetics and Safety After a Single Dose of Imarikiren in Subjects with Renal or Hepatic Impairment. Clin Drug Investig. 2018 Nov;38(11):1041-1051. doi: 10.1007/s40261-018-0695-4. PMID 30194585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Japan from 1 March 2015 to 10 June 2016.
Pre-assignment Details: Participants with normal renal (1R) and hepatic (1H) function; those who had historical diagnosis of renal (mild [2R], moderate [3R], severe or end-stage renal failure with no hemodialysis [4R], end-stage renal failure [with hemodialysis] [5R]); hepatic impairment (mild [2H] and moderate [3H]) were enrolled to receive TAK-272 40 milligram (mg).
Groups:
- Cohort 1R: Normal Renal Function: Participants with normal renal function (estimated glomerular filtration rate [eGFR] greater than or equal to [>=] 90 milliliter per minute per 1.73 square meter [mL/min/1.73 m^2]) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period.
- Cohort 2R: Mild Renal Impairment: Participants with mild renal impairment (eGFR >=60, less than [<] 90 mL/min/1.73 m^2) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period.
- Cohort 3R: Moderate Renal Impairment: Participants with moderate renal impairment (eGFR >=30, <60 mL/min/1.73 m^2) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period.
- Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis): Participants with severe or end-stage renal failure undergoing no hemodialysis (eGFR <30 mL/min/1.73 m^2) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period.
- Cohort 5R: End-stage Renal Failure (Hemodialysis): Participants with hemodialysis received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period in Part 1 (dialysis on Day 1 after dosing). After Part 1 follow-up period, then the same participants received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period in Part 2 (non-dialysis on Day 1). Participants who completed Cohort 5R-Part 1 started Part 2 after completion of 2-day of follow up in Part 1.
- Cohort 1H: Normal Hepatic Function: Participants with normal hepatic function received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period.
- Cohort 2H: Mild Hepatic Impairment: Participants with mild hepatic impairment (Child-Pugh class A score of 5-6) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period. The Child-Pugh classification assesses the severity of 5 hepatic parameters (total serum bilirubin, serum albumin, prothrombin time [PT] or prothrombin time international normalized ratio [INR], ascites and encephalopathy grade) on a scale of 1 (none) to 3 (moderate). Total hepatic impairment score ranges from 5 (mild) to 15 (severe) where higher score indicates more severity.
- Cohort 3H: Moderate Hepatic Impairment: Participants with moderate hepatic impairment (Child-Pugh class B score of 7-9) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period. The Child-Pugh classification assesses the severity of 5 hepatic parameters (total serum bilirubin, serum albumin, PT or INR, ascites and encephalopathy grade) on a scale of 1 (none) to 3 (moderate). Total hepatic impairment score ranges from 5 (mild) to 15 (severe) where higher score indicates more severity.
Period: Overall Study
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The plasma pharmacokinetic (PK) set included all participants treated with the study drug who had no significant protocol deviation, satisfied the minimum protocol provisions, and could be evaluated for plasma PK.
Groups:
- Cohort 1R: Normal Renal Function: Participants with normal renal function (eGFR>=90 mL/min/1.73 m^2) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period.
- Cohort 2R: Mild Renal Impairment: Participants with mild renal impairment (eGFR >=60,< 90 mL/min/1.73 m^2) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period.
- Cohort 2H: Mild Hepatic Impairment: Participants with mild hepatic impairment (Child-Pugh class A score of 5-6) received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period. The Child-Pugh classification assesses the severity of 5 hepatic parameters (total serum bilirubin, serum albumin, PT or INR, ascites and encephalopathy grade) on a scale of 1 (none) to 3 (moderate). Total hepatic impairment score ranges from 5 (mild) to 15 (severe) where higher score indicates more severity.
- Total: Total of all reporting groups
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (5.61) | 59.7 (8.94) | 70.2 (5.53) | 69.5 (5.89) | 71.2 (6.91) | 61.0 (5.73) | 61.0 (10.41) | 61.5 (8.96) | 65.0 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 1 | 3 | 2 | 2 | 14
  Male | 3 | 5 | 5 | 5 | 5 | 3 | 4 | 4 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 157.3 (10.91) | 163.7 (9.18) | 167.7 (5.32) | 159.0 (8.63) | 160.8 (5.56) | 161.2 (5.64) | 160.0 (10.20) | 161.5 (11.40) | 161.4 (8.54)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 57.58 (6.328) | 59.80 (11.726) | 69.87 (5.654) | 56.48 (9.392) | 60.83 (6.982) | 62.25 (6.275) | 65.08 (11.760) | 69.73 (23.171) | 62.70 (11.674)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.42 (2.807) | 22.12 (2.289) | 24.88 (2.082) | 22.22 (2.588) | 23.62 (3.242) | 24.03 (2.935) | 25.33 (3.389) | 26.03 (5.581) | 23.96 (3.303)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 2 | 4 | 3 | 2 | 3 | 2 | 3 | 1 | 20
  Current smoker | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 4 | 10
  Ex-smoker | 4 | 1 | 1 | 4 | 2 | 3 | 2 | 1 | 18
Alcohol Classification [Count of Participants; unit: Participants]
  Drinks every day | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 6
  Drinks a few days per week | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 9
  Drinks a few days per month | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 7
  Never drinks | 2 | 2 | 4 | 3 | 5 | 2 | 4 | 4 | 26
Caffeine Classification [Count of Participants; unit: Participants] — Participants who were answered Yes or No for a question "Take Caffeine in Daily Life?" were reported.
  Participants
    Yes | 5 | 6 | 5 | 6 | 5 | 6 | 3 | 2 | 38
    No | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 4 | 10
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 114.8 (26.03) | 80.7 (17.70) | 54.8 (9.50) | 16.3 (7.61) | 4.5 (0.55) | 115.2 (14.55) | 93.7 (21.63) | 100.8 (16.49) | 72.6 (43.41)
Alpha1 Acid Glycoprotein (AGP) [Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)] | 64.97 (12.065) | 48.65 (4.809) | 70.30 (14.936) | 114.45 (25.029) | 82.77 (7.104) | 55.80 (17.694) | 51.18 (16.328) | 41.12 (20.282) | 66.15 (26.757)

OUTCOME MEASURES:

1. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Free Form of TAK-272 (TAK-272F) and Its Metabolite M-I
Time Frame: Day 1: Pre-dose and at multiple time points (0.5, 1, 1.5, 2, 3, 4, 5, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120 hours post dose; up to 120 hours) post-dose
Population: The plasma PK set included all participants treated with the study drug who had no significant protocol deviation, satisfied the minimum protocol provisions, and could be evaluated for plasma PK.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis): Part 1 is hemodialysis part in the Cohort 5R. Participants with hemodialysis received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period in Part 1 (hemodialysis on Day 1 after dosing).
- Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis): Part 2 is non-hemodialysis part in the Cohort 5R. Participants with hemodialysis received TAK-272 40 mg, tablets, orally in fasted state, once on Day 1 of a 6-day treatment period with 2-day follow-up period in Part 2 (non-hemodialysis on Day 1). Participants who completed Cohort 5R-Part 1 started Part 2 after completion of 2-day follow up period in Part 1.
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL)
  TAK-272F | 2951 (391.70) | 1507 (952.72) | 3481 (797.67) | 8053 (2964.7) | 4579 (1091.2) | 5409 (1343.0) | 2269 (366.43) | 2307 (750.08) | 3085 (1551.3)
  M-I | 50.66 (27.097) | 31.58 (13.765) | 47.22 (18.319) | 138.9 (89.619) | 104.3 (20.684) | 132.3 (40.166) | 33.95 (13.432) | 38.18 (14.860) | 60.01 (27.427)
Statistical Analysis 1: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; TAK-272F: Least square mean (LS) mean cohort ratios for the test groups (Cohort 2R) and the reference group (Cohort 1R) with their 95 percent (%) confidence intervals (CI) were calculated using an analysis of variance (ANOVA) model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 51.08, 95% CI 2-sided [35.22 to 74.08]
Statistical Analysis 2: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; TAK-272F: LS mean cohort ratios for the test groups (Cohort 3R) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 117.95, 95% CI 2-sided [81.32 to 171.07]
Statistical Analysis 3: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); TAK-272F: LS mean cohort ratios for the test groups (Cohort 4R) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 272.87, 95% CI 2-sided [188.14 to 395.76]
Statistical Analysis 4: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); TAK-272F: LS mean cohort ratios for the test groups (Cohort 5R-Part 2) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 183.27, 95% CI 2-sided [126.36 to 265.81]
Statistical Analysis 5: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; TAK-272F: LS mean cohort ratios for the test groups (Cohort 2H) and the reference group (Cohort 1H) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 101.67, 95% CI 2-sided [68.95 to 149.90]
Statistical Analysis 6: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; TAK-272F: LS mean cohort ratios for the test groups (Cohort 3H) and the reference group (Cohort 1H) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 135.98, 95% CI 2-sided [92.23 to 200.50]
Statistical Analysis 7: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; M-I: LS mean cohort ratios for the test groups (Cohort 2R) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 62.34, 95% CI 2-sided [36.17 to 107.45]
Statistical Analysis 8: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; M-I: LS mean cohort ratios for the test groups (Cohort 3R) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 93.20, 95% CI 2-sided [54.08 to 160.64]
Statistical Analysis 9: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); M-I: LS mean cohort ratios for the test groups (Cohort 4R) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 274.21, 95% CI 2-sided [159.10 to 472.63]
Statistical Analysis 10: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); M-I: LS mean cohort ratios for the test groups (Cohort 5R-Part 2) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 261.12, 95% CI 2-sided [151.50 to 450.05]
Statistical Analysis 11: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; M-I: LS mean cohort ratios for the test groups (Cohort 2H) and the reference group (Cohort 1H) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 112.47, 95% CI 2-sided [69.34 to 182.41]
Statistical Analysis 12: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; M-I: LS mean cohort ratios for the test groups (Cohort 3H) and the reference group (Cohort 1H) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 176.75, 95% CI 2-sided [108.97 to 286.67]

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-272F and Its Metabolite M-I
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  TAK-272F | 753.5 (211.81) | 432.2 (248.57) | 580.5 (312.90) | 1555 (303.45) | 1061 (222.54) | 1078 (417.38) | 522.8 (111.65) | 446.0 (198.78) | 688.1 (339.69)
  M-I | 20.08 (11.909) | 14.13 (7.0952) | 11.05 (7.9919) | 25.30 (13.442) | 19.86 (5.6056) | 20.87 (3.5431) | 12.45 (8.8158) | 11.45 (6.2582) | 17.34 (6.6026)
Statistical Analysis 1: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; TAK-272F: LS mean cohort ratios for the test groups (Cohort 2R) and the reference group (Cohort 1R) with their 95% CIs were calculated using an ANOVA model for natural log-transformed data; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 57.36, 95% CI 2-sided [37.76 to 87.14]
Statistical Analysis 2: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 77.04, 95% CI 2-sided [50.72 to 117.03]
Statistical Analysis 3: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 206.41, 95% CI 2-sided [135.88 to 313.54]
Statistical Analysis 4: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 143.11, 95% CI 2-sided [94.21 to 217.39]
Statistical Analysis 5: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 85.31, 95% CI 2-sided [51.03 to 142.61]
Statistical Analysis 6: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 131.63, 95% CI 2-sided [78.74 to 220.04]
Statistical Analysis 7: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 70.38, 95% CI 2-sided [40.42 to 122.53]
Statistical Analysis 8: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 55.03, 95% CI 2-sided [31.61 to 95.81]
Statistical Analysis 9: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 125.96, 95% CI 2-sided [72.35 to 219.30]
Statistical Analysis 10: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 103.93, 95% CI 2-sided [59.70 to 180.95]
Statistical Analysis 11: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 91.97, 95% CI 2-sided [49.45 to 171.06]
Statistical Analysis 12: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 139.33, 95% CI 2-sided [74.91 to 259.15]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-272F and Its Metabolite M-I
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL
  TAK-272F | 2971 (393.33) | 1527 (953.59) | 3519 (812.10) | 8106 (3004.0) | 4647 (1101.8) | 5471 (1342.1) | 2289 (368.39) | 2326 (746.40) | 3126 (1575.2)
  M-I | 62.32 (32.579) | 36.87 (15.778) | 60.47 (21.246) | 162.0 (99.759) | 129.6 (23.022) | 198.8 (95.110) | 38.84 (15.615) | 50.52 (16.916) | 74.82 (31.470)
Statistical Analysis 1: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 51.39, 95% CI 2-sided [35.45 to 74.49]
Statistical Analysis 2: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 118.43, 95% CI 2-sided [81.70 to 171.68]
Statistical Analysis 3: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 272.83, 95% CI 2-sided [188.21 to 395.50]
Statistical Analysis 4: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 184.13, 95% CI 2-sided [127.02 to 266.91]
Statistical Analysis 5: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 101.64, 95% CI 2-sided [69.04 to 149.64]
Statistical Analysis 6: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 136.59, 95% CI 2-sided [92.78 to 201.09]
Statistical Analysis 7: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 59.17, 95% CI 2-sided [33.99 to 102.99]
Statistical Analysis 8: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 97.04, 95% CI 2-sided [55.75 to 168.90]
Statistical Analysis 9: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 260.03, 95% CI 2-sided [149.39 to 452.60]
Statistical Analysis 10: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 319.06, 95% CI 2-sided [183.31 to 555.34]
Statistical Analysis 11: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 130.07, 95% CI 2-sided [81.66 to 207.18]
Statistical Analysis 12: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 192.63, 95% CI 2-sided [120.94 to 306.83]

4. Primary Outcome: AUClast,u: Area Under the Unbound Plasma Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration for TAK-272F
Description: AUClast,u is the area under the concentration-time curve of the unbound drug in plasma over the time interval from 0 to time of last quantifiable post-dose of TAK-272.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 138.7 (72.422) | 83.51 (40.288) | 135.0 (16.105) | 154.7 (55.009) | 162.9 (40.127) | 192.4 (55.731) | 107.7 (17.583) | 145.5 (82.297) | 348.5 (102.16)
Statistical Analysis 1: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 60.22, 95% CI 2-sided [40.05 to 90.56]
Statistical Analysis 2: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 97.39, 95% CI 2-sided [64.77 to 146.46]
Statistical Analysis 3: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 111.60, 95% CI 2-sided [74.21 to 167.82]
Statistical Analysis 4: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 138.79, 95% CI 2-sided [92.29 to 208.70]
Statistical Analysis 5: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 135.18, 95% CI 2-sided [87.91 to 207.87]
Statistical Analysis 6: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 323.75, 95% CI 2-sided [210.54 to 497.85]

5. Primary Outcome: Cmax,u: Maximum Unbound Plasma Concentration for TAK-272F
Description: Cmax,u is the peak unbound plasma concentration of a drug after administration, obtained directly from the unbound plasma concentration-time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 35.38 (20.053) | 23.92 (12.222) | 22.54 (10.180) | 29.88 (5.8353) | 37.76 (11.566) | 38.41 (22.002) | 24.82 (7.1225) | 28.11 (17.659) | 77.66 (23.421)
Statistical Analysis 1: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 67.61, 95% CI 2-sided [42.17 to 108.39]
Statistical Analysis 2: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 63.70, 95% CI 2-sided [39.73 to 102.12]
Statistical Analysis 3: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 84.45, 95% CI 2-sided [52.67 to 135.38]
Statistical Analysis 4: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 108.54, 95% CI 2-sided [67.70 to 174.01]
Statistical Analysis 5: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 113.25, 95% CI 2-sided [69.62 to 184.24]
Statistical Analysis 6: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 312.89, 95% CI 2-sided [192.34 to 509.00]

6. Primary Outcome: AUC∞,u: Area Under the Unbound Plasma Concentration-time Curve From Time 0 to Infinity for TAK-272F
Description: AUC∞,u is the area under the concentration-time curve of the unbound drug in plasma over the time interval from 0 to infinity of TAK-272.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 139.3 (73.070) | 84.51 (40.355) | 136.5 (16.537) | 155.5 (56.099) | 165.1 (39.885) | 194.6 (55.238) | 108.5 (17.885) | 146.5 (82.800) | 352.9 (103.09)
Statistical Analysis 1: Comparison: Cohort 1R: Normal Renal Function vs Cohort 2R: Mild Renal Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 60.68, 95% CI 2-sided [40.35 to 91.27]
Statistical Analysis 2: Comparison: Cohort 1R: Normal Renal Function vs Cohort 3R: Moderate Renal Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 98.01, 95% CI 2-sided [65.17 to 147.41]
Statistical Analysis 3: Comparison: Cohort 1R: Normal Renal Function vs Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 111.68, 95% CI 2-sided [74.25 to 167.96]
Statistical Analysis 4: Comparison: Cohort 1R: Normal Renal Function vs Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 139.70, 95% CI 2-sided [92.88 to 210.11]
Statistical Analysis 5: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 2H: Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 135.08, 95% CI 2-sided [87.75 to 207.92]
Statistical Analysis 6: Comparison: Cohort 1H: Normal Hepatic Function vs Cohort 3H: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; LS Mean Cohort Ratio (%) = 325.28, 95% CI 2-sided [211.32 to 500.70]

7. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-272F and Its Metabolite M-I
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hour
  TAK-272F | 0.7500 [0.500 to 1.50] | 0.5000 [0.500 to 1.50] | 1.000 [0.500 to 3.00] | 1.000 [0.500 to 1.50] | 0.7250 [0.417 to 0.950] | 0.9815 [0.450 to 1.43] | 1.000 [0.500 to 1.00] | 0.5170 [0.500 to 1.00] | 0.5000 [0.500 to 0.500]
  M-I | 0.7500 [0.500 to 1.00] | 0.7500 [0.500 to 1.50] | 0.7500 [0.500 to 1.50] | 1.000 [0.500 to 1.50] | 0.7250 [0.417 to 0.950] | 0.9250 [0.450 to 1.42] | 1.000 [0.500 to 1.00] | 1.000 [0.500 to 1.00] | 0.5000 [0.500 to 1.00]

8. Primary Outcome: Apparent Clearance (CL/F) for TAK-272F
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
liter per hour (L/hr) | 13.57 (1.8565) [0.500 to 1.50] | 28.05 (9.3870) [0.500 to 1.50] | 11.63 (2.6246) [0.500 to 3.00] | 5.290 (2.3246) [0.500 to 1.50] | 8.955 (3.0987) | 7.535 (2.1430) | 17.68 (3.1682) | 17.83 (5.0433) | 13.70 (5.1084)

9. Primary Outcome: CLu/F: Apparent Clearance for Unbound Drug After Extravascular Administration for TAK-272F
Description: CLu/F is the apparent clearance for unbound drug after extravascular administration of TAK-272.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/hr | 315.7 (152.20) [0.500 to 1.00] | 500.8 (163.96) [0.500 to 1.50] | 294.7 (34.938) [0.500 to 1.50] | 271.5 (100.55) [0.500 to 1.50] | 247.8 (60.579) | 210.2 (46.940) | 372.8 (66.949) | 301.8 (139.68) | 117.3 (33.417)

10. Primary Outcome: Cumulative Urinary Excretion Ratio of TAK-272F and Its Metabolite M-I From 0 to 72 Hours Post-dose in Cohorts 1R, 2R, 3R, 4R, 1H, 2H and 3H
Description: Urinary excretion ratio (percentage [%] of dose) of TAK-272 and its metabolite M-I in urine was calculated for each participant.
Time Frame: Day 1: Pre-dose and at multiple time points (4, 8, 12, 24, 36, 48, 72 hours post dose; up to 72 hours) post-dose
Population: The urine PK analysis population where urinary excretion data on Day 1 was available. The urine PK set included all participants treated with the study drug who had no significant protocol deviation, satisfied the minimum protocol provisions, and could be evaluated for urine PK.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
percentage of dose
  TAK-272F | 13.227 (1.3321) | 10.710 (3.2216) | 12.820 (2.6621) | 4.947 (3.3152) | 13.980 (5.0380) | 15.205 (2.6194) | 21.222 (4.9429)
  M-I | 0.558 (0.2596) | 0.477 (0.2017) | 0.284 (0.0598) | 0.072 (0.0462) | 0.453 (0.1515) | 0.557 (0.1672) | 0.788 (0.3352)

11. Primary Outcome: Plasma Protein Binding Rate of TAK-272F in Cohorts 1R, 2R, 3R, 4R, 5R, 1H, 2H and 3H
Description: Plasma protein binding rate was the percentage of unbound fraction of TAK-272F in plasma protein.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of unbound fraction of TAK-272F
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
% of unbound fraction of TAK-272F | 5.298 (3.1279) | 5.597 (0.88260) | 3.970 (0.88091) | 1.948 (0.35549) | 3.598 (0.59734) | 4.800 (0.77095) | 7.177 (4.0484) | 12.82 (6.5481)

12. Primary Outcome: Excretion Ratio of TAK-272F in Dialysate in Cohort 5R
Description: Excretion ratio (% of dose) of TAK-272F in dialysis fluid was calculated for each participant.
Time Frame: Day 1: Pre-dose, up to 6 hours post-dose
Population: The dialysate PK set included all participants treated with the study drug who had no significant protocol deviation, satisfied the minimum protocol provisions, and could be evaluated for dialysate PK.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis)
Number analyzed (Participants) | 6
percentage of dose | 3.110 (0.8911)

13. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE)
Time Frame: Baseline up to Day 8 of each Cohort
Population: The safety analysis set included all participants who were treated with at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 3

14. Secondary Outcome: Number of Participants With TEAE Related to Vital Signs
Description: Number of participants with TEAE related to vital signs was reported in this outcome measure. The related event to report was only "Blood Pressure Decreased" throughout this study.
Time Frame: Baseline up to Day 8 of each Cohort
Population: The safety analysis set included all participants who were treated with at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1

15. Secondary Outcome: Number of Participants With TEAE Related to Body Weight
Description: Number of participants with TEAE related to body weight was reported in this outcome measure. There were no events to report as TEAE related to body weight throughout this study.
Time Frame: Baseline up to Day 8 of each Cohort
Population: The safety analysis set included all participants who were treated with at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With TEAE Related to 12-lead Electrocardiograms (ECG)
Description: Number of participants with TEAE related to ECG was reported in this outcome measure. There were no events to report as TEAE related to ECG throughout this study.
Time Frame: Baseline up to Day 8 of each Cohort
Population: The safety analysis set included all participants who were treated with at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With TEAE Related to Laboratory Tests
Description: Number of participants with TEAE related to laboratory tests was reported in this outcome measure. The related event to report was only "Alanine Aminotransferase Increased" throughout this study.
Time Frame: Baseline up to Day 8 of each Cohort
Population: The safety analysis set included all participants who were treated with at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to Day 8 of each Cohort
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1R: Normal Renal Function | Cohort 2R: Mild Renal Impairment | Cohort 3R: Moderate Renal Impairment | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) | Cohort 1H: Normal Hepatic Function | Cohort 2H: Mild Hepatic Impairment | Cohort 3H: Moderate Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/6 | 2/6 | 2/6 | 1/6 | 1/6 | 1/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1R: Normal Renal Function (N=6) | Cohort 2R: Mild Renal Impairment (N=6) | Cohort 3R: Moderate Renal Impairment (N=6) | Cohort 4R: Severe or End-stage Renal Failure(Non-hemodialysis) (N=6) | Cohort 5R-Part 1: End-stage Renal Failure (Hemodialysis) (N=6) | Cohort 5R-Part 2: End-stage Renal Failure (Hemodialysis) (N=6) | Cohort 1H: Normal Hepatic Function (N=6) | Cohort 2H: Mild Hepatic Impairment (N=6) | Cohort 3H: Moderate Hepatic Impairment (N=6)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dumping syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.